CLINICAL TRIAL: NCT07240272
Title: Modulation of Executive Functions and Speech in Parkinson's Disease by Theta tACS Targeted at the Medial Frontal Cortex
Brief Title: tACS Modulates Speech and Cognitive Impairments in People With PD by Targeting the Medial Frontal Cortex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ke Dong, MD (Other)
Responsible Party: Sponsor-Investigator, Ke Dong, MD, Research Associate, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nos.82172528
Record Dates: First submitted 2025-09-26; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; transcranial alternating current stimulation; medial frontal cortex; executive functions; speech disorder
MeSH Terms: conditions — Parkinson Disease; Speech Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6Hz-group (Experimental)
  Interventions: Other: 6Hz-tACS
- Sham-group (Sham Comparator)
  Interventions: Other: Sham-tACS

INTERVENTIONS:
Other: 6Hz-tACS — tACS applied to the MFC at a frequency of 6 Hz, using a high-definition 1×4 electrode configuration with individualized current intensity, delivered for 20 minutes.
  Arms: 6Hz-group
Other: Sham-tACS — Except for turning down the current intensity to zero during the 20-minute period, all other parameters are identical to those in 6Hz-group.
  Arms: Sham-group

SUMMARY:
This clinical trial aims to study whether transcranial alternating current stimulation (tACS) applied to the medial frontal cortex (MFC) can improve speech and cognitive function in people with Parkinson's disease (PD), and to evaluate the safety of tACS. The main goals are to answer the following questions:

1. Can tACS stimulation of the MFC improve executive functions in people with PD (such as reasoning, planning, inhibition, and complex problem-solving)?
2. Can it improve the integration of auditory information and speech motor control during communication?

Researchers will compare the effects of real tACS versus sham (placebo) stimulation to see if real stimulation leads to better speech and cognitive outcomes in PD patients.

Participants will:

1. Receive one extra 20-minute session of either real or sham tACS each day for two weeks
2. Attend clinic visits before stimulation, right after the 2-week period, and again at 1 month and 3 months for assessments and tests
3. Have their executive function scores, speech performance, and related brain activity recorded

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Parkinson's disease.
2. Aged 35-80 years.
3. Absence of non-PD neurological disorders.
4. No hearing impairment, dementia, psychiatric abnormalities, or history of neurosurgical treatment.

Exclusion Criteria:

1. Pregnancy.
2. Any contraindications to electrical stimulation.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Verbal Fluency Test (VFT) | Assessments were completed at baseline, after two weeks of stimulation, and at 1- and 3-month follow-ups.
  The VFT assesses abilities such as thought initiation, rapid word retrieval, and cognitive flexibility. It has two parts: 1.Phonemic Fluency Test (PFT), people needed to name as many Chinese words as possible beginning with "fa" or "xiao" within 60 seconds. 2.Semantic Fluency Test (SFT), people needed to name as many items as possible from categories such as "fruits," "vegetables," "animals," and "occupations" within 60 seconds. The number of correct and non-repeated words produced within the time limit were recorded.
Digit Span Test (DST) | Assessments were completed at baseline, after two weeks of stimulation, and at 1- and 3-month follow-ups.
  The DST assesses working memory and selective attention. People repeat a series of numbers in the same order (forward) or reverse order (backward) as spoken by the examiner. The maximum correctly repeated sequence length was recorded.
Trail Making Test (TMT) | Assessments were completed at baseline, after two weeks of stimulation, and at 1- and 3-month follow-ups.
  The TMT assesses complex visual scanning, conceptual tracking, cognitive flexibility and divided attention. It has two parts: TMT-A: People draw a trail by connecting 25 Arabic numbers in ascending order. TMT-B: the trail alternates between connecting 12 Arabic numbers and 12 Chinese characters. The time taken to complete each task is recorded.
Speech motor integration ability as assessed by a well-established paradigm: frequency-altered feedback (FAF) task | Assessments were completed at baseline, after two weeks of stimulation, and at 1- and 3-month follow-ups.
  In the FAF task, participants needed to sit in a sound-attenuated room and produce the vowel /u/ according to instructions. The acoustic signal is recorded and randomly shifted in pitch by an external device. The pitch-shifted voice is then fed back to the participant. This unexpected pitch perturbation elicits either an opposite or a following acoustic compensation response. The amplitude and timing of this response are recorded and used to assess the participant's speech-motor integration ability.

OTHER OUTCOMES:
The event-related potentials (ERPs) components recorded by Electroencephalography (EEG) | Assessments were completed at baseline, after two weeks of stimulation, and at 1- and 3-month follow-ups.
  During the FAF task, cortical electrical activity associated with the pitch perturbation event was simultaneously recorded. Using the perturbation onset as the zero point, a time window ranging from -500ms to 700ms was defined. The peak amplitude and latency of N1 and P2 components were extracted within 80-180 ms and 160-280 ms time windows after the perturbation onset, respectively.
The hemodynamic responses in the executive process as assessed by Functional Near-Infrared Spectroscopy (fNIRS) | Assessments were completed at baseline, after two weeks of stimulation, and at 1- and 3-month follow-ups.
  The fNIRS monitoring was conducted during a VFT task consisting of multiple 30-second blocks. The average change in oxygenated hemoglobin concentration during the task was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation Medicine, The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code